CLINICAL TRIAL: NCT04186260
Title: A Gender and Culturally Specific Approach to Reduce NAFLD in Mexican-American Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1911187047; KMD014761A (Other Grant/Funding Number: NIMHD)
Record Dates: First submitted 2019-11-27; First posted 2019-12-04 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: NAFLD
Keywords: obesity; overweight; Mexican; Mexican-American; men; weight loss
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Overweight; Multiple Endocrine Neoplasia Type 1; Weight Loss

STUDY DESIGN:
Intervention Model Description: The pilot study uses a small randomized-controlled trial (RCT) design that will be conducted in two phases. The first phase includes recruitment, screening, and baseline assessment procedures. The second phase will include PNPLA3 risk allele carriers (CG/GG genotype) with NAFLD, who will be assigned 2:1 to a NAFLD-specific weight loss intervention tailored for Mexican-American men, including informing them of their lifestyle and genetic risk, for 12-months compared to a wait-list control group.
Who Masked: Outcomes Assessor
Masking Description: Assessments will be performed at 0, 6, and 12-months post-intervention. To minimize the potential for bias, outcome assessors will be blinded to treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAFLD-specific weight loss intervention (Experimental): Participants will attend 12 weekly 30-45-minute individual counseling sessions and receive tailored lesson materials focused on behavioral strategies for adopting and maintaining healthy eating and physical activity (PA) behaviors. Participants will self-monitor their body weight, eating, and PA behaviors in a weekly journal. Dietary recommendations will follow nutritional guidelines for the treatment of NAFLD. To facilitate the adoption of the dietary recommendation, participants will be provided culturally-tailored meal plans and grocery lists that allow them to make small, practical dietary changes of ~100 calories. Participants will be prescribed weekly exercise goals with the duration increasing from 15-45 minutes, 5 days/week, over the 12-month program. After the completion of 12 weekly individual counseling sessions, participants will complete a 12-week follow-up including bi-weekly phone calls, followed by a 6-month follow-up period in which no intervention contact is made.
  Interventions: Behavioral: NAFLD-specific weight loss intervention
- Wait-list control (Other): The wait-list control group will receive the same intervention strategies described for the NAFLD-specific weight loss intervention after study comparisons have been made.
  Interventions: Other: Wait-list control

INTERVENTIONS:
Behavioral: NAFLD-specific weight loss intervention — This is a 12-month NAFLD-specific weight loss intervention that is explicitly tailored for Mexican-American men. It will include recommendations for diet, physical activity, and will utilize risk for NAFLD as a mechanism to engage men in lifestyle modification.
  Arms: NAFLD-specific weight loss intervention
Other: Wait-list control — Participants in this condition will not receive treatment for 12-months until study comparisons have been made. After 12-months, participants will receive the 12-month NAFLD-specific weight loss intervention.
  Arms: Wait-list control

SUMMARY:
Using a small Randomized Controlled Trial (RCT) study design, PNPLA3 risk allele carriers (CG/GG genotype) with NAFLD, will be assigned 2:1 to a tailored NAFLD-specific weight loss intervention compared to a wait-list control group.

DETAILED DESCRIPTION:
The Mexican-American population accounts for 64.3% of the U.S. Hispanic population and is the fastest growing Hispanic subgroup. Non-alcoholic fatty liver disease (NAFLD) is a chronic disease associated with obesity that is highest in the nation for Mexican-American men. NAFLD consists of a spectrum of conditions, ranging from fatty liver to cirrhosis and liver cancer. Lack of physical activity and sugar-sweetened beverage consumption are risk factors for NAFLD and are highly evident in the Mexican-American male population. Additionally, Mexican-American men are at increased risk of NAFLD and liver cancer if they are carriers of a version of a gene (PNPLA3) found to increase risk and severity of NAFLD. In the absence of prescription medications, weight loss due to changes in diet and physical activity is recommended for the prevention and treatment of NAFLD. Changes in lifestyle that result in >5% body weight loss have been shown to improve levels of liver fat and even reverse the condition. Despite the clear need to develop effective intervention strategies for Mexican-American men, no studies to date have explored the use of health risk assessment strategies, including genetic risk, to motivate behavior change to reduce the risk of NAFLD in Mexican-American men. Consequently, this will be the first weight loss intervention for Mexican-American men to incorporate genetic predisposition and lifestyle risk factors of NAFLD (e.g., dietary sugar consumption), as a strategy to improve engagement in weight loss and weight maintenance behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as a Mexican or Mexican-American man
* 18-64 years of age
* BMI between 30 to 50.0 kg/m²
* Have a CAP score ≥248 at screening
* Be identified as PNPLA3 risk allele carriers (CG/GG genotype) at screening
* Be able to provide informed consent
* Speak, read, and write either English and/or Spanish.

Exclusion Criteria:

* Have active, chronic gastrointestinal disorder (e.g. inflammatory bowel disease, ulcerative colitis, Chron's disease, celiac disease)
* Been previously diagnosed with viral hepatitis, liver disease or liver cancer
* Have a history of bariatric surgery
* Report medical condition or treatment for a medical condition that could affect body weight or ability to engage in structured physical activity that is consistent with the intervention for this study
* Have current congestive heart failure, angina, uncontrolled arrhythmia, or other symptoms indicative of an increased acute risk for a cardiovascular event
* Have a resting systolic blood pressure of ≥150 mmHg or resting diastolic blood pressure of ≥100 mmHg
* Have an eating disorders that would contraindicate weight loss or physical activity
* Report significant alcohol consumption (e.g., drinking ≥ 21 standard drinks/week, binge drinkers, or those with previous heavy alcohol consumption) identified by the Alcohol Use Disorders Identification Test
* Currently treated for psychological issues (e.g., depression, bipolar disorder, etc.), taking psychotropic medications with the previous 12 months, or hospitalized for depression within the previous 5 years
* Report exercise on ≥3 days per week for ≥ 20 minutes per day over the past 3 months
* Report weight loss of ≥5% or participating in a weight reduction diet program in the past 3 months
* Taking any medication or supplement known to affect body composition or history of exposure to hepatotoxic drugs
* Report plans to relocate to a location that limits their access to the study site or having employment, personal, or travel commitments that prohibit attendance to all of the scheduled assessments.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Study Recruitment: Interest in Participation at Baseline | Baseline
  The number of Mexican-American men who express interest in participation.
Study Recruitment: Screened for Eligibility at Baseline | Baseline
  The number of Mexican-American men screened for eligibility.
Study Recruitment: Eligibility at Baseline | Baseline
  The number of Mexican-American men eligible/ineligible for study inclusion and reason for ineligibility.
Study Recruitment: Enrollment at Baseline | Baseline
  The number of Mexican-American men enrolled in the study.
Retention at 6-months | 6-months
  Retention will be measured as the number of participants who remain in the study at 6-months, divided by the number enrolled.
Retention at 12-months | 12-months
  Retention will be measured as the number of participants who remain in the study at 12-months, divided by the number enrolled.
Attendance at weekly counseling sessions at 6-months | 6-months
  The investigators will use descriptive analyses to examine attendance at weekly counseling sessions (% sessions attended) at 6-months.
Attendance at weekly counseling sessions at 12-months | 12-months
  The investigators will use descriptive analyses to examine attendance at weekly counseling sessions (% sessions attended) at 12-months.
Self-monitoring of dietary intake at 6-months | 6-months
  The investigators will use descriptive analyses to examine self-monitoring of dietary intake (% days completed) at 6-months.
Self-monitoring of dietary intake at 12-months | 12-months
  The investigators will use descriptive analyses to examine self-monitoring of dietary intake (% days completed) at 12-months.
Self-monitoring of physical activity at 6-months | 6-months
  The investigators will use descriptive analyses to examine self-monitoring of physical activity (% days completed) at 6-months.
Self-monitoring of physical activity at 12-months | 12-months
  The investigators will use descriptive analyses to examine self-monitoring of physical activity (% days completed) at 12-months.
Self-weighing behaviors at 6-months | 6-months
  The investigators will use descriptive analyses to examine self-weighing behaviors (average days/week) at 6-months.
Self-weighing behaviors at 12-months | 12-months
  The investigators will use descriptive analyses to examine self-weighing behaviors (average days/week) at 12-months.
Intervention delivery time at 6-months | 6-months
  The investigators will use descriptive analyses to examine intervention delivery time (average minutes/week) at 6-months.
Intervention delivery time at 12-months | 12-months
  The investigators will use descriptive analyses to examine intervention delivery time (average minutes/week) at 12-months.
Treatment Satisfaction at 6-months: rating | 6-months
  Participants will be asked to rate their overall satisfaction (Treatment Satisfaction Survey; Minimum Score: 1 = very dissatisfied and Maximum Score: 4 = very satisfied) with the tailored weight loss intervention at 6-months.
Treatment Satisfaction at 12-months: rating | 12-months
  Participants will be asked to rate their overall satisfaction (Treatment Satisfaction Survey; Minimum Score: 1 = very dissatisfied and Maximum Score: 4 = very satisfied) with the tailored weight loss intervention at 12-months.

SECONDARY OUTCOMES:
Change in body weight at 6-months | 6-months
  Body weight (kg) will be measured on a digital scale to assess change in body weight at 6-months over the intervention period.
Change in body weight at 12-months | 12-months
  Body weight (kg) will be measured on a digital scale to assess change in body weight at 12-months over the intervention period.
Change in waist circumference at 6-months | 6-months
  Waist circumference (cm) will be assessed using a standardized protocol at 6-months.
Change in waist circumference at 12-months | 12-months
  Waist circumference (cm) will be assessed using a standardized protocol at 12-months.
Change in liver steatosis at 6-months | 6-months
  A non-invasive transient elastography (FibroScan®, TE) will be used to measure the amount of fat (steatosis) present in the liver at 6-months based on controlled attenuation parameters (CAP).
Change in liver steatosis at 12-months | 12-months
  A non-invasive transient elastography (FibroScan®, TE) will be used to measure the amount of fat (steatosis) present in the liver at 12-months based on controlled attenuation parameters (CAP).
Change in liver fibrosis at 6-months | 6-months
  A non-invasive transient elastography (FibroScan®, TE) will be used to measure the amount of liver fibrosis (scaring) present in the liver at 6-months based on kilopascals (kPa).
Change in liver fibrosis at 12-months | 12-months
  A non-invasive transient elastography (FibroScan®, TE) will be used to measure the amount of liver fibrosis (scaring) present in the liver at 12-months based on kilopascals (kPa).
Change in alanine aminotransferase (ALT) at 6-months | 6-months
  Fasting blood samples will be collected to examine changes in alanine aminotransferase (ALT) in Units/Liter (U/L) at 6-months.
Change in alanine aminotransferase (ALT) at 12-months | 12-months
  Fasting blood samples will be collected to examine changes in alanine aminotransferase (ALT) in Units/Liter (U/L) at 12-months.
Change in aspartate aminotransferase (AST) at 6-months | 6-months
  Fasting blood samples will be collected to examine changes in aspartate aminotransferase (AST) in Units/Liter (U/L) at 6-months.
Change in aspartate aminotransferase (AST) at 12-months | 12-months
  Fasting blood samples will be collected to examine changes in aspartate aminotransferase (AST) in Units/Liter (U/L) at 12-months.
Change in physical activity at 6-months | 6-months
  An Actigraph will be used to objectively measure and quantify energy expenditure from physical activity at 6-months.
Change in physical activity at 12-months | 12-months
  An Actigraph will be used to objectively measure and quantify energy expenditure from physical activity at 12-months.
Change in dietary intake at 6-months | 6-months
  24-hr recalls will be used to assess self reported food intake (kcal/day) at 6-months. This will be used to estimate calories, dietary fat, protein, and carbohydrates consumed.
Change in dietary intake at 12-months | 12-months
  24-hr recalls will be used to assess self reported food intake (kcal/day) at 12-months. This will be used to estimate calories, dietary fat, protein, and carbohydrates consumed.
Change in weight loss self-efficacy at 6-months: questionnaire | 6-months
  Change in weight loss self-efficacy at 6-months will be measured using a reliable and validated self reported questionnaire (Weight Efficacy Lifestyle Questionnaire; 10-point Likert scale from 0 (not confident) to 9 (very confident)).
Change in weight loss self-efficacy at 12-months: questionnaire | 12-months
  Change in weight loss self-efficacy at 12-months will be measured using a reliable and validated self reported questionnaire (Weight Efficacy Lifestyle Questionnaire; 10-point Likert scale from 0 (not confident) to 9 (very confident)).

CONTACTS AND LOCATIONS:
Overall Officials: David O Garcia, PhD, Principal Investigator — University of Arizona, Mel & Enid Zuckerman College of Public Health
Locations (1):
- University of Arizona Collaboratory for Metabolic Disease Prevention and Treatment, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will be stripped of identifiers prior to release for sharing. Dr. Garcia will make the data and associated documentation available to users under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. The final dataset, including all study variables, will be developed for import into standard statistical software programs including SPSS, SASS and STATA.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The final dataset will be cleaned and organized during the final study year and will be available only to the study PI or designees (Co-Investigators, Collaborators) for 36-months post-study completion. At that time the dataset then will be made more widely available through data use agreements with the PI/University of Arizona. Access will require registration including investigator name, credentials, and academic affiliation.
Access Criteria: Dr. Garcia will make the data and associated documentation available to users under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. All study data collection forms will be made available as pdf files; data collection time-points and dictionary of data definitions also will be made available.

REFERENCES:
- [Background] Kallwitz ER, Daviglus ML, Allison MA, Emory KT, Zhao L, Kuniholm MH, Chen J, Gouskova N, Pirzada A, Talavera GA, Youngblood ME, Cotler SJ. Prevalence of suspected nonalcoholic fatty liver disease in Hispanic/Latino individuals differs by heritage. Clin Gastroenterol Hepatol. 2015 Mar;13(3):569-76. doi: 10.1016/j.cgh.2014.08.037. Epub 2014 Sep 15. PMID 25218670
- [Background] Lazo M, Bilal U, Perez-Escamilla R. Epidemiology of NAFLD and Type 2 Diabetes: Health Disparities Among Persons of Hispanic Origin. Curr Diab Rep. 2015 Dec;15(12):116. doi: 10.1007/s11892-015-0674-6. PMID 26468154
- [Background] Saab S, Manne V, Nieto J, Schwimmer JB, Chalasani NP. Nonalcoholic Fatty Liver Disease in Latinos. Clin Gastroenterol Hepatol. 2016 Jan;14(1):5-12; quiz e9-10. doi: 10.1016/j.cgh.2015.05.001. Epub 2015 May 11. PMID 25976180
- [Background] Romeo S, Kozlitina J, Xing C, Pertsemlidis A, Cox D, Pennacchio LA, Boerwinkle E, Cohen JC, Hobbs HH. Genetic variation in PNPLA3 confers susceptibility to nonalcoholic fatty liver disease. Nat Genet. 2008 Dec;40(12):1461-5. doi: 10.1038/ng.257. Epub 2008 Sep 25. PMID 18820647
- [Background] Severson TJ, Besur S, Bonkovsky HL. Genetic factors that affect nonalcoholic fatty liver disease: A systematic clinical review. World J Gastroenterol. 2016 Aug 7;22(29):6742-56. doi: 10.3748/wjg.v22.i29.6742. PMID 27547017
- [Background] Tilg H, Moschen A. Weight loss: cornerstone in the treatment of non-alcoholic fatty liver disease. Minerva Gastroenterol Dietol. 2010 Jun;56(2):159-67. PMID 20485253
- [Background] Martinez LA, Larrieta E, Kershenobich D, Torre A. The Expression of PNPLA3 Polymorphism could be the Key for Severe Liver Disease in NAFLD in Hispanic Population. Ann Hepatol. 2017 November-December,;16(6):909-915. doi: 10.5604/01.3001.0010.5282. PMID 29055919
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2985-3023. doi: 10.1016/j.jacc.2013.11.004. Epub 2013 Nov 12. No abstract available. PMID 24239920
- [Background] Musso G, Cassader M, Rosina F, Gambino R. Impact of current treatments on liver disease, glucose metabolism and cardiovascular risk in non-alcoholic fatty liver disease (NAFLD): a systematic review and meta-analysis of randomised trials. Diabetologia. 2012 Apr;55(4):885-904. doi: 10.1007/s00125-011-2446-4. Epub 2012 Jan 27. PMID 22278337